CLINICAL TRIAL: NCT00005212
Title: Work Organization and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1091; R29HL039633 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine the combined effects of job strain and social isolation on cardiovascular morbidity and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Much of the medical and epidemiological research on the causes of cardiovascular disease has concentrated either on individual life style behaviors such as smoking and exercise or on biomedical risk factors such as hypertension, and diabetes. This research has provided the basis for improvements in personal health behaviors and in the treatment of hypertension which has reduced the incidence of cardiovascular disease in this country. However, even the best statistical models, incorporating all such risk factors, leave a significant proportion of cardiovascular disease mortality and morbidity unexplained. Major differences in cardiovascular disease rates have also been observed between different social classes and different societies. These findings have led epidemiologists and sociomedical researchers to investigate other types of variables, including psychosocial factors, such as personal predispositions, social support networks, and work-related stress. A series of studies, in a variety of disciplines, suggested that occupational stress may contribute to the development of cardiovascular disease.

A major source of data was the Swedish Survey of Living Conditions (ULF). The ULF was drawn from a sample which included the total occupational and demographic variation of an entire society. The survey contained information on age, sex, marital status, occupational class background and nationality of respondents and parents, residence, education, past employment history and income data.

DESIGN NARRATIVE:

In this non-concurrent prospective study, ten years of follow-up data were linked with five years of data from the Survey of Living Conditions collected between 1976 and 1980. Total and cause-specific mortality data were obtained from the Swedish National Death Registry and morbidity incidence data from the Registry of Hospitalizations. The relationship between the duration of exposure time and disease risk was examined utilizing occupational history information which was combined with Theorell's Occupational Psychosocial Scoring System. Logistic regression analysis was used to examine the relative risks associated with adverse work characteristics and to test for potential interactions and confounding effects. Cox's proportional hazards model was used as an approximation of life table methods. Analysis was performed separately for men and women.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-03; Study Completion 1993-02 (Actual)

REFERENCES:
- [Background] Johnson JV, Hall EM. Job strain, work place social support, and cardiovascular disease: a cross-sectional study of a random sample of the Swedish working population. Am J Public Health. 1988 Oct;78(10):1336-42. doi: 10.2105/ajph.78.10.1336. PMID 3421392
- [Background] Johnson JV, Hall EM, Theorell T. Combined effects of job strain and social isolation on cardiovascular disease morbidity and mortality in a random sample of the Swedish male working population. Scand J Work Environ Health. 1989 Aug;15(4):271-9. doi: 10.5271/sjweh.1852. PMID 2772582
- [Background] Johnson JV, Hall EM: Social Support in the Work Environment and Cardiovascular Disease. In: Shumaker S, Czajkowski S (Eds.), Social Support and Cardiovascular Disease. New York: Plenum Press, in press, 1988
- [Background] Johnson JV: Control, Collectively and the Psychosocial Work Environment. In: Sauter S, Hurrell J, Cooper C (Eds), Job Stress and Work Control. New York: Academic Press, in press, 1988
- [Background] Johansson G, Johnson JV, Hall EM. Smoking and sedentary behavior as related to work organization. Soc Sci Med. 1991;32(7):837-46. doi: 10.1016/0277-9536(91)90310-9. PMID 2028279
- [Background] Hall EM, Johnson JV, Tsou TS. Women, occupation, and risk of cardiovascular morbidity and mortality. Occup Med. 1993 Oct-Dec;8(4):709-19. PMID 8303487
- [Background] Johnson JV, Stewart WF. Measuring work organization exposure over the life course with a job-exposure matrix. Scand J Work Environ Health. 1993 Feb;19(1):21-8. doi: 10.5271/sjweh.1508. PMID 8465168